CLINICAL TRIAL: NCT05388903
Title: A Phase 1, Subjects- and Investigator-Blinded, Sponsor-Unblinded, Placebo-Controlled, Randomized, Sequential Cohort Study to Assess the Safety and Pharmacokinetics of Single Ascending Subcutaneous and Intravenous Doses of DS-2325a in Healthy Subjects
Brief Title: A Study to Assess the Safety and Pharmacokinetics of Single Ascending Subcutaneous and Intravenous Doses of DS-2325a in Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Daiichi Sankyo (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Double | Purpose: Treatment
Other Study IDs: DS2325-104
Record Dates: First submitted 2022-05-19; First posted 2022-05-24 (Actual); Last update posted 2023-03-06 (Actual); Status verified 2023-03

CONDITIONS: Netherton Syndrome
Keywords: Netherton Syndrome; DS-2325a; Healthy Participants
MeSH Terms: conditions — Netherton Syndrome

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- DS-2325a SC (Experimental): Participants who will be randomized to receive DS-2325a as a fixed dose subcutaneous (SC) injection (starting dose 30 mg).
  Interventions: Drug: DS-2325a
- Placebo SC (Placebo Comparator): Participants who will be randomized to receive placebo as a subcutaneous (SC) injection.
  Interventions: Drug: Placebo
- DS-2325a IV (Experimental): Participants who will be randomized to receive DS-2325a as a fixed dose intravenous (IV) infusion (starting dose 100 mg).
  Interventions: Drug: DS-2325a
- Placebo IV (Placebo Comparator): Participants who will be randomized to receive placebo as an intravenous infusion.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: DS-2325a — Subcutaneous injection (starting dose 30 mg)
  Arms: DS-2325a SC
Drug: DS-2325a — Intravenous infusion (starting dose 100 mg)
  Arms: DS-2325a IV
Drug: Placebo — Subcutaneous injection
  Arms: Placebo SC
Drug: Placebo — Intravenous infusion
  Arms: Placebo IV

SUMMARY:
Netherton syndrome (NS) is a rare autosomal recessive disease and no systemic treatment or standard of care currently exists for patients with NS. DS-2325a, a specific and potent inhibitor of kallikrein 5, is expected to treat NS by replacing a defective gene.

DETAILED DESCRIPTION:
This first-in-human study for DS-2325a will evaluate the safety, tolerability, and pharmacokinetics of single ascending doses of DS-2325a in healthy participants. DS-2325a will be evaluated after both subcutaneous (SC) injections and intravenous (IV) infusions, as it may have to be given intravenously to young patients and as loading dose.

ELIGIBILITY:
Inclusion Criteria:

* Participants must give written informed consent to participation in the study prior to Screening
* Healthy men and women 18 to 45 years of age (inclusive), with a BMI of 18 kg/m2 to 30 kg/m^2 (inclusive) at Screening
* All women must have a negative serum pregnancy test at Screening and all women of childbearing potential must have a negative urine pregnancy test on Day -1
* Women must not be lactating during the study treatment period and for 3 months after the last dose of study treatment
* Women of childbearing potential must practice effective contraception during the study treatment period and for 3 months after the last dose of study treatment. They must agree to use 2 different means of nonhormonal contraceptive methods
* Women of non-childbearing potential must be either surgically sterile (ie, bilateral tubal ligation at least 3 months prior to dosing) or in menopausal state confirmed as follows: 1 year of spontaneous amenorrhea without an alternative medical cause and a serum FSH level ≥40 mIU/mL
* Men must agree to use contraception (condom with spermicide) during the study treatment period and for at least 3 months after the last dose of study treatment or be surgically sterile (vasectomy at least 3 months prior to dosing)
* Women should not donate eggs and men should not donate sperm during the study treatment period and for at least 3 months after the last dose of study treatment
* Participants must be in good health as determined by Screening medical history, physical examination, vital signs, ECGs, serum chemistry, hematology, virology, and urinalysis performed at Screening and on Day -1

Exclusion Criteria:

* History or current chronic lung disease including asthma, chronic obstructive pulmonary disease (COPD), or heavy smoking of >10 pack years
* Previous or current treatment with systemic corticosteroids or any immunosuppressive agents
* Participants who have received a transfusion or any blood products within the last year prior to dosing
* Participants who have made any blood donation or have had a loss of blood of ≥500 mL within 56 days prior to the dose of study drug
* Participants who consume more than 21 units of alcohol per week (1 unit of alcohol equals 1/2 pint of beer, 4 ounces of wine, or 1 ounce of spirits) or those participants who have a significant history of alcoholism or drug/chemical abuse within the last 2 years.
* Participants with positive results on tests for drugs of abuse, cotinine, or alcohol at Screening and/or Day -1.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 64 (Actual)
Dates: Start 2022-06-20 (Actual); Primary Completion 2023-01-26 (Actual); Study Completion 2023-01-26 (Actual)

PRIMARY OUTCOMES:
Number of Participants with Any Treatment-emergent Adverse Events Following Administration of DS-2325a | Screening (Day -28 to -3) pre-dose up to Day 57 post-dose
  Treatment-emergent adverse events (TEAEs) are defined as new adverse events (AEs) that occur after the dose of study drug or as AEs that were present prior to the dose of study drug but which worsened in severity after the start of study drug.

SECONDARY OUTCOMES:
Pharmacokinetic Parameter Area Under the Concentration Curve (AUC) | SC and IV cohorts: Day 1 pre-dose and 1, 2, 4, 8 hours (hr) post-dose; 24, 48, 96, 120, 144, 168, 192, 240, 288, 336, 384, 432, 480, 552, 624, 696, 768, 840, 1008, 1176, 1344 hr post-dose
  Pharmacokinetic parameters will be calculated for DS-2325a by noncompartmental methods.
Pharmacokinetic Parameter Time to Maximum Concentration (Tmax) | SC and IV cohorts: Day 1 pre-dose and 1, 2, 4, 8 hours (hr) post-dose; 24, 48, 96, 120, 144, 168, 192, 240, 288, 336, 384, 432, 480, 552, 624, 696, 768, 840, 1008, 1176, 1344 hr post-dose
  Pharmacokinetic parameters will be calculated for DS-2325a by noncompartmental methods.
Pharmacokinetic Parameter Maximum Concentration (Cmax) | SC and IV cohorts: Day 1 pre-dose and 1, 2, 4, 8 hours (hr) post-dose; 24, 48, 96, 120, 144, 168, 192, 240, 288, 336, 384, 432, 480, 552, 624, 696, 768, 840, 1008, 1176, 1344 hr post-dose
  Pharmacokinetic parameters will be calculated for DS-2325a by noncompartmental methods.
Pharmacokinetic Parameter Last Measurable Time (Tlast) | SC and IV cohorts: Day 1 pre-dose and 1, 2, 4, 8 hours (hr) post-dose; 24, 48, 96, 120, 144, 168, 192, 240, 288, 336, 384, 432, 480, 552, 624, 696, 768, 840, 1008, 1176, 1344 hr post-dose
  Pharmacokinetic parameters will be calculated for DS-2325a by noncompartmental methods.
Pharmacokinetic Parameter Elimination Rate Constant Associated With the Terminal Phase (Kel) | SC and IV cohorts: Day 1 pre-dose and 1, 2, 4, 8 hours (hr) post-dose; 24, 48, 96, 120, 144, 168, 192, 240, 288, 336, 384, 432, 480, 552, 624, 696, 768, 840, 1008, 1176, 1344 hr post-dose
  Pharmacokinetic parameters will be calculated for DS-2325a by noncompartmental methods.
Pharmacokinetic Parameter Elimination Half-life (T1/2) | SC and IV cohorts: Day 1 pre-dose and 1, 2, 4, 8 hours (hr) post-dose; 24, 48, 96, 120, 144, 168, 192, 240, 288, 336, 384, 432, 480, 552, 624, 696, 768, 840, 1008, 1176, 1344 hr post-dose
  Pharmacokinetic parameters will be calculated for DS-2325a by noncompartmental methods.
Number of Participants Who Are Anti-Drug Antibody (ADA)-Positive (Baseline and Post-Baseline) and Number of Participants Who Have Treatment-emergent ADA | Day 1 pre-dose and 336 hours (hr), 552 hrs, 696 hrs, and 1344 hrs post-dose
  Blood samples will be collected to determine ADAs.

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Director, Study Director — Daiichi Sankyo
Locations (1):
- Worldwide Clinical Trials, San Antonio, Texas, United States

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participant data (IPD) on completed studies and applicable supporting clinical trial documents may be available upon request at https://vivli.org/. In cases where clinical trial data and supporting documents are provided pursuant to our company policies and procedures, Daiichi Sankyo will continue to protect the privacy of our clinical trial participants. Details on data sharing criteria and the procedure for requesting access can be found at this web address: https://vivli.org/ourmember/daiichi-sankyo/
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Completed studies that has reached a global end or completion with all data set collected and analyzed, and for which the medicine and indication have received European Union (EU) and United States (US), and/or Japan (JP) marketing approval on or after 01 January 2014 or by the US or EU or JP Health Authorities when regulatory submissions in all regions are not planned and after the primary study results have been accepted for publication.
Access Criteria: Formal request from qualified scientific and medical researchers on IPD and clinical study documents on completed clinical trials supporting products submitted and licensed in the United States, the European Union and/or Japan from 01 January 2014 and beyond for the purpose of conducting legitimate research. This must be consistent with the principle of safeguarding study participants' privacy and consistent with provision of informed consent.
URL: https://vivli.org/ourmember/daiichi-sankyo/